CLINICAL TRIAL: NCT06373705
Title: Utilizing a Multi-Physics Cardiac Simulator for Surgical Planning in Complex Congenital Heart Disease Pediatric Patients
Brief Title: Cardiac Simulator for Surgical Planning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alison Lesley Marsden, DOUGLASS M. AND NOLA LEISHMAN PROFESSOR OF CARDIOVASCULAR DISEASES, PROFESSOR OF PEDIATRICS (CARDIOLOGY) AND OF BIOENGINEERING AND, BY COURTESY, OF MECHANICAL ENGINEERING, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 74566; 1R01HL173845-01 (NIH)
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Congenital Heart Disease in Children

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to either receive standard of care "on the fly" surgical planning discussion as is current practice or assisted surgical planning discussion with the aid of computer simulation.
Masking Description: After consent to participate in the study, patient will be entered into a random allocation sequence for standard of care (SOC) or cardiac simulator groups.
  Patient and surgeon will both be notified which group they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgical planning discussion without cardiac simulator (No Intervention): Conventional surgical planning discussion without cardiac simulator
- Surgical planning discussion with aid of cardiac simulator (Experimental): Surgical planning discussion with aid of cardiac simulator
  Interventions: Device: Cardiac simulator

INTERVENTIONS:
Device: Cardiac simulator — A computer software cardiac simulator for surgical planning in complex Congenital Heart Disease (CHD) pediatric patients.
  Arms: Surgical planning discussion with aid of cardiac simulator

SUMMARY:
The goal of this clinical trial is to learn if a computer software program (cardiac simulator) for surgical planning will lead to improvements in patient care by decreasing the incidence of unsuccessful interventions and reinterventions for pediatric patients with congenital heart disease. It is not a commercially available device to treat congenital heart disease in pediatric patients. The main aims are:

To provide safe pre-operative testing of surgical approaches with a computer model cardiac simulator.

To aid surgeons in envisioning different surgical approaches for each individual patient.

To bolster the standard of care surgical planning discussions which will be particularly useful for patients with unique, complex congenital heart disease.

Participants will:

Consent to being randomized with a 50% chance of receiving standard of care "on the fly" surgical planning discussion as is current practice or assisted surgical planning discussion with the aid of the computer software cardiac simulator.

Receive results of their computer simulated findings during their surgical planning discussion if they are in the cardiac simulator group.

DETAILED DESCRIPTION:
The computer software will be developed at the Cardiovascular Biomechanics Computation Lab at Stanford.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are pediatric patients ages 0-17 with a congenital heart disease (CHD) diagnosis of 1) congenitally corrected transposition of the great arteries (cc-TGA) with ventricular septal defect (VSD), 2) double outlet right ventricle (DORV) with remote VSD, or 3) other single ventricle conditions.

Exclusion Criteria:

* Adult patients with CHD.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Mortality | At date of hospital discharge or up to 30 days post-operation
  Alive or deceased post-operative

SECONDARY OUTCOMES:
Mortality | Latest follow-up exam up to 3 years post-operation
  Alive or deceased long-term
Number of cardioplegic arrest | Up to 10 hours
  Due to quality of pathways to blood flow, function of inlet and outlet valves, or residual hemodynamic lesions during operation (up to 5 times)

OTHER OUTCOMES:
Number of repair revisions needed | At date of hospital discharge or up to 30 days post-operation
  Due to quality of pathways to blood flow, function of inlet and outlet valves, residual hemodynamic lesions
Time on cardiopulmonary bypass | Up to approximately 10 hours intra-operation
  Hours and minutes of operative duration
Ventricular function | Immediately post-operation, at date of discharge, follow-up to 3 years
  Echocardiogram
Ventricular function | At 1 year post-operation
  MRI
Ventricular function | At 1 year post-operation
  Catheterization
Valvular function | Immediately post-operation, at date of discharge, follow-up to 3 years
  Echocardiogram
Valvular function | At 1 year post-operation
  MRI
Valvular function | Valvular function
  Catheterization
Number of days in hospital post-operation | At discharge date up to 180 days
  Length of time from date of operation to discharge from hospital
Type of post-operative inotrope | At discharge date up to approximately 3 weeks
  What inotropes were administered post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Alison Marsden, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No